CLINICAL TRIAL: NCT01111448
Title: Treatment of MDS Patients With Single Agent Temsirolimus - a Pilot Study
Brief Title: Temsirolimus in Myelodysplastic Syndrome (MDS)
Acronym: TEMDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unfavourable Risk-Benefit-Ratio
Sponsor: Technische Universität Dresden (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-TEMDS1-042
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndromes of all IPSS subgroups
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus (Experimental): 25 mg/day 1; 8; 15; 22 of each 28-day cycle
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — 25 mg/day 1; 8; 15; 22 of each 28-day cycle as intravenous infusion over 30 min

SUMMARY:
The goal of this Pilot-study is to evaluate the response of unselected MDS patients to temsirolimus a drug approved for the treatment of renal cell cancer. It is planned to give temsirolimus at a weekly dose of 25 mg as intravenous infusion for a maximum duration of 12 months. Regular bone marrow biopsies are planned for controlling MDS response.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at the time of signing the informed consent form;
* Patients able to understand the consequences of participating in this trial and not having any disorders or other circumstances (i.e. being in ward or imprisoned) which keeps them from giving written informed consent;
* cytologically or histologically established diagnosis of de novo or therapy-related MDS according to the FAB-classification, either previously treated or untreated, presenting with:

  * Group I (low-risk): Low- or INT-1 risk features according to IPSS and requiring at least 4 units of red blood cells within the last 8 weeks prior to screening visit or presenting with neutropenia (<1 Gpt/l neutrophils) or
  * Group II (high-risk): INT-2 or HIGH-risk IPSS refractory or intolerant to 5-Azacytidine.

CMML patients of dysplastic phenotype (WBC < 13 Gpt/l) may be included in both arms according to IPSS. CMML patients showing proliferative phenotype (WBC >=13 Gpt/l) will be included in the high risk arm;

* not eligible for an immediate allogeneic HSCT or conventional chemotherapy;
* all previous MDS specific therapies (except supportive approaches like transfusions or antibiotics) must have been discontinued at least 4 weeks prior to study enrollment;
* ECOG performance status of <= 3 at study entry;
* laboratory test results within these ranges:

  * Serum creatinine <= 177 µmo/l (<= 2.0 mg/dL);
  * total bilirubin <= 3 x ULN;
  * AST (SGOT) and ALT (SGPT) <= 3 x ULN;
  * total fasting cholesterol <= 9.1 mmol/l (350 mg/dl);
  * fasting triglyceride level <= 4.5 mmol/l (400 mg/dl);
  * platelets > 25 Gpt/l without transfusion support in patients with LOW- and INT-1 Risk according to IPSS;
* signed informed consent.

Exclusion Criteria:

* For Patients with LOW- or INT1-Risk according to IPSS: Thrombocytopenia below 25 Gpt/l (INT2- and HIGH-IPSS patients may be included irrespective of platelet count);
* known hypersensitivity to temsirolimus, sirolimus or any components of the infusion solution (dl-alpha-tocopherol, propylene glycol, anhydrous citric acid, polysorbate 80, polyethylene glycol 400, dehydrated alcohol);
* known hypersensitivity to macrolid antibiotics (because of structural similarities between this class of antibiotics and study medication);
* any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study;
* known positive for HIV or any other uncontrolled infection;
* presence of any other malignancy being not in complete remission for at least 3 years (previous chemotherapy for other malignancies is not an exclusion criteria);
* necessity of therapeutic anticoagulation (excluding low dose ASS);
* participation in an other clinical trial within the last 4 weeks;
* pregnant or breast feeding females (lactating females must agree not to breast feed while on study);
* females of childbearing potential (FCBP) except those fulfilling at least one of the following criteria:

  * post-menopausal (12 months of natural amenorrhea or 6 months of amenorrhea with serum FSH > 40 U/ml);
  * post-surgery (6 weeks after bilateral ovarectomy with or without hysterectomy);regular and correct use of contraceptives with a PEARL Index of < 1% (e.g. implants, depot formulations of hormones, oral contraceptives, intra uterine device - IUD);
  * sexual abstinence;
  * partner, who had vasectomy (confirmed by two negative analyses of semen);
* male patients, who do not agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 3 months following discontinuation from the study even if he has undergone a successful vasectomy;
* patients with a history of chronic drug abuse or another illness which does not allow the patient to assess the nature and/or possible consequences of the study;
* patients who are not likely to follow the trial protocol (lack of willingness to cooperate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Overall hematological response rate using modified IWG criteria (combination of CR, PR, marrow-CR and SD with HI). | at 4 months

SECONDARY OUTCOMES:
Toxicity as measured by NCI CTCAE v3.0 | 4 and 12 months
Overall survival | 1 year
Progression-free-survival | 1 year
Rate of leukemic progression | 1 year
Overall hematological response rate using modified IWG-criteria | 1 year
Quality of life as measured by EORTC-QLQ30 | 4 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, MD, PhD, Principal Investigator — Medizinische Klinik I, Universitätsklinikum Carl-Gustav-Carus, Dresden, Germany
Locations (7):
- Germany (7):
  - Klinikum Chemnitz Klinik für Innere Medizin III, Chemnitz
  - Universitätsklinikum C. G. Carus der TU Dresden, Dresden
  - Universitätsklinikum Düsseldorf Klinik für Hämatologie, Onkologie und Klin. Immunologie, Düsseldorf
  - Universitätsmedizin Göttingen Georg-August-Universität Abteilung Hämatologie und Onkologie, Göttingen
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Forschungsgesellschaft mbH, Leipzig
  - Klinikum Mannheim GmbH III. Medizinische Universitätsklinik -SP Hämatologie/Onkologie, Mannheim